CLINICAL TRIAL: NCT06108752
Title: Comparative Effect of Scapular Stabilization Versus Thoracic Extension Exercises on Pain, Disability, Range of Motion, and Craniovertebral Angle in Young Adults With Text Neck Syndrome.
Brief Title: Comparative Effect of Scapular Stabilization vs Thoracic Extension Exercises in Young Adults With Text Neck Syndrome.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0161
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Neck Syndrome; Forward Head Posture
Keywords: Craniovertebral angle; Scapular stabilization exercises; Thoracic extension; Text neck syndrome; Range of motion; Pain; Disability
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scapular Stabilization Exercises (Experimental): Scapular stabilization exercises along with the hot pack and cervical active range of motion exercises
  Interventions: Other: Scapular stabilization exercises
- Thoracic Extension Exercises (Experimental): Thoracic extension exercises along with the hot pack and cervical active range of motion exercises
  Interventions: Other: Thoracic extension exercises

INTERVENTIONS:
Other: Scapular stabilization exercises — The scapular stabilization exercises will be comprised of four exercise programs. Each exercise will be performed with two sets of 15 reps, 10 sec per rep 40 min per day, thrice per week for a total of six weeks. Baseline treatment will be the application of a hot pack for 7-10 minutes and cervical active range of motion exercises.
  Arms: Scapular Stabilization Exercises
Other: Thoracic extension exercises — Thoracic extension exercises will be comprised of three exercise programs. Each exercise will be performed with two sets of 15 reps, 10 sec per rep 40 min per day, thrice per week for a total of six weeks. Baseline treatment will be the application of a hot pack for 7-10 minutes and cervical active range of motion exercises.
  Arms: Thoracic Extension Exercises

SUMMARY:
The aim of the study is to compare the effect of scapular stabilization versus thoracic extension exercises on pain, disability, range of motion, and cranio-vertebral angle in young adults with Text Neck Syndrome.

DETAILED DESCRIPTION:
Text neck has emerged as a widespread modern epidemic that affects people of all ages, particularly younger populations, as they are exposed to handheld mobile device use for several hours a day beginning at a very early age. The relation between the posture due to handheld mobile device use and neck pain is still debatable. To manage the maladaptive posture of the cervical spine, indirect treatment instead of direct treatment of the neck can be used, which is the basis for the concept of regional interdependence, i.e., the cause of pain becomes the cause of damage to other body parts. Therefore, not treating the damaged part, but indirectly treating the area of cause can alleviate the symptoms. A bio-dynamic relationship between the cervical and thoracic spine is associated with exercise, an important factor causing neck pain. Therefore, many clinicians pay attention to the thoracic spine of patients with neck pain and recommend thoracic extension exercises. On the other hand, many researchers recommended scapular stabilization exercise as a recovery treatment for imbalanced scapular muscles caused by forward head posture.

This study investigates how exercise programs not directly applied to the cervical spine affect people with text neck syndrome. The significance of the current study is to evaluate the comparison between concentric and eccentric exercise which is previously rarely investigated.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female participants with forward head posture or text neck syndrome
* Participants with neck pain from the past three months
* Smart-phones must be used for at least ≥3 hours each day
* Participants with craniovertebral angle <53° will be included in this study

Exclusion Criteria:

* History of cervical and thoracic spine surgery within the past three months
* Serious pathological conditions within the past three months
* Congenital spinal anomalies, or rheumatoid arthritis
* Neurological signs and severe psychological disorders

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-12-08 (Estimated); Study Completion 2024-01-08 (Estimated)

PRIMARY OUTCOMES:
Neck disability index (NDI) | 6 weeks
  Changes from baseline. NDI is a valid and reliable tool having values ranging from 0.50 to 0.98.
  The NDI assessment involves a 10-item, 50-point index questionnaire that assesses the effects of neck pain and symptoms during a range of functional activities.
Visual analogue scale (VAS) | 6 weeks
  Changes from baseline. The visual analogue scale (VAS) is a simple and frequently used method for the assessment of variations in intensity of pain. The reliability of the VAS for disability is moderate to good i.e. 0.98. However, its validity is questionable.
Goniometer for cervical range of motion | 6 weeks
  Changes from baseline. Goniometer has fair inter-tester reliability ranging from 0.79-0.92. Validity of this tool is good i.e. 0.97-0.98 This tool is most commonly used in the clinical settings for evaluating joint range of motion.
Photogrammetry for craniovertebral angle (image j software) | 6 weeks
  Changes from baseline. 'Image J', is an analysis software with high reliability and validity.
  This study will assess the craniovertebral angle using a digital camera. The camera will be placed 1.5 m from the participant's right side to take a lateral photographic view of the participant's head and neck in a seated position. The craniovertebral angle is the angle between the horizontal line passing the 7th Cervical vertebra (C7) and the line extending from C7 to the tragus of the ear. The resulting maladaptive posture of the neck will be determined using Image J software.

CONTACTS AND LOCATIONS:
Overall Officials: Faiza Amjad, M.Phil, Principal Investigator — Riphah International University
Locations (1):
- Punjab Employees Social Security Institute, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kang NY, Im SC, Kim K. Effects of a combination of scapular stabilization and thoracic extension exercises for office workers with forward head posture on the craniovertebral angle, respiration, pain, and disability: A randomized-controlled trial. Turk J Phys Med Rehabil. 2021 Sep 1;67(3):291-299. doi: 10.5606/tftrd.2021.6397. eCollection 2021 Sep. PMID 34870115
- [Background] Warda DG, Nwakibu U, Nourbakhsh A. Neck and Upper Extremity Musculoskeletal Symptoms Secondary to Maladaptive Postures Caused by Cell Phones and Backpacks in School-Aged Children and Adolescents. Healthcare (Basel). 2023 Mar 10;11(6):819. doi: 10.3390/healthcare11060819. PMID 36981476
- [Background] Cho J, Lee E, Lee S. Upper thoracic spine mobilization and mobility exercise versus upper cervical spine mobilization and stabilization exercise in individuals with forward head posture: a randomized clinical trial. BMC Musculoskelet Disord. 2017 Dec 12;18(1):525. doi: 10.1186/s12891-017-1889-2. PMID 29233164
- [Background] Kong YS, Kim YM, Shim JM. The effect of modified cervical exercise on smartphone users with forward head posture. J Phys Ther Sci. 2017 Feb;29(2):328-331. doi: 10.1589/jpts.29.328. Epub 2017 Feb 24. PMID 28265167
- [Background] Fiebert I, Kistner F, Gissendanner C, DaSilva C. Text neck: An adverse postural phenomenon. Work. 2021;69(4):1261-1270. doi: 10.3233/WOR-213547. PMID 34366308
- [Background] Koseki T, Kakizaki F, Hayashi S, Nishida N, Itoh M. Effect of forward head posture on thoracic shape and respiratory function. J Phys Ther Sci. 2019 Jan;31(1):63-68. doi: 10.1589/jpts.31.63. Epub 2019 Jan 10. PMID 30774207
- [Background] Singla D, Veqar Z. Association Between Forward Head, Rounded Shoulders, and Increased Thoracic Kyphosis: A Review of the Literature. J Chiropr Med. 2017 Sep;16(3):220-229. doi: 10.1016/j.jcm.2017.03.004. Epub 2017 Sep 28. PMID 29097952
- [Background] Moezy A, Sepehrifar S, Solaymani Dodaran M. The effects of scapular stabilization based exercise therapy on pain, posture, flexibility and shoulder mobility in patients with shoulder impingement syndrome: a controlled randomized clinical trial. Med J Islam Repub Iran. 2014 Aug 27;28:87. eCollection 2014. PMID 25664288
- [Background] Yoo WG. Effect of thoracic stretching, thoracic extension exercise and exercises for cervical and scapular posture on thoracic kyphosis angle and upper thoracic pain. J Phys Ther Sci. 2013 Nov;25(11):1509-10. doi: 10.1589/jpts.25.1509. Epub 2013 Dec 11. PMID 24396221
- [Background] Alpayci M, Ilter S. Isometric Exercise for the Cervical Extensors Can Help Restore Physiological Lordosis and Reduce Neck Pain: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2017 Sep;96(9):621-626. doi: 10.1097/PHM.0000000000000698. PMID 28118272
- [Background] Suvarnnato T, Puntumetakul R, Uthaikhup S, Boucaut R. Effect of specific deep cervical muscle exercises on functional disability, pain intensity, craniovertebral angle, and neck-muscle strength in chronic mechanical neck pain: a randomized controlled trial. J Pain Res. 2019 Mar 7;12:915-925. doi: 10.2147/JPR.S190125. eCollection 2019. PMID 30881101
- [Background] Ghamkhar L, Arab AM, Nourbakhsh MR, Kahlaee AH, Zolfaghari R. Examination of Regional Interdependence Theory in Chronic Neck Pain: Interpretations from Correlation of Strength Measures in Cervical and Pain-Free Regions. Pain Med. 2020 Feb 1;21(2):e182-e190. doi: 10.1093/pm/pnz206. PMID 31504861
- [Background] Suwaidi ASA, Moustafa IM, Kim M, Oakley PA, Harrison DE. A Comparison of Two Forward Head Posture Corrective Approaches in Elderly with Chronic Non-Specific Neck Pain: A Randomized Controlled Study. J Clin Med. 2023 Jan 9;12(2):542. doi: 10.3390/jcm12020542. PMID 36675471
- [Background] Nejati P, Lotfian S, Moezy A, Moezy A, Nejati M. The relationship of forward head posture and rounded shoulders with neck pain in Iranian office workers. Med J Islam Repub Iran. 2014 May 3;28:26. eCollection 2014. PMID 25250268
- [Background] Sindhu BS, Shechtman O, Tuckey L. Validity, reliability, and responsiveness of a digital version of the visual analog scale. J Hand Ther. 2011 Oct-Dec;24(4):356-63; quiz 364. doi: 10.1016/j.jht.2011.06.003. Epub 2011 Aug 6. PMID 21820864
- [Background] Dindaroglu F, Kutlu P, Duran GS, Gorgulu S, Aslan E. Accuracy and reliability of 3D stereophotogrammetry: A comparison to direct anthropometry and 2D photogrammetry. Angle Orthod. 2016 May;86(3):487-94. doi: 10.2319/041415-244.1. Epub 2015 Aug 12. PMID 26267357
- [Background] Dissanayaka TD, Pallegama RW, Suraweera HJ, Johnson MI, Kariyawasam AP. Comparison of the Effectiveness of Transcutaneous Electrical Nerve Stimulation and Interferential Therapy on the Upper Trapezius in Myofascial Pain Syndrome: A Randomized Controlled Study. Am J Phys Med Rehabil. 2016 Sep;95(9):663-72. doi: 10.1097/PHM.0000000000000461. PMID 26945216